CLINICAL TRIAL: NCT06603519
Title: Determining the Impact of Dietary Intervention on Inflammation and Microbiome Composition in Patients With Recurrent Polyps Post-Colonoscopy.
Brief Title: Impact of Dietary Intervention on Inflammation and Microbiome Composition Post-Colonoscopy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Seerave Foundation (Unknown)
Responsible Party: Principal Investigator, Jack Gilbert, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 809457
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Polyp; Inflammation; Dietary Intervention; Microbiota; Colorectal Neoplasms; Metabolomics
Keywords: Dietary Intervention; Inflammation; Microbiome; Polyps; Colonoscopy; Gut Health; Nutrition; Human Microbiome; Fecal Metabolomics; Serum Metabolomics; Metabolomics Analysis
MeSH Terms: conditions — Inflammation; Colorectal Neoplasms; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention Group (Experimental): Participants in this arm will follow a modified plant-based Mediterranean diet following their colonoscopies. The dietary intervention aims to reduce inflammation and improve gut microbiome composition. Participants' gut bacteria and overall health will be monitored through blood and stool sample collections, focusing on inflammation reduction and metabolic health improvement.
  Interventions: Dietary Supplement: Modified Plant-Based Mediterranean Diet

INTERVENTIONS:
Dietary Supplement: Modified Plant-Based Mediterranean Diet — Two-week dietary intervention after the participants' scheduled colonoscopy consisting of vegetarian high-fiber meals. These meals are designed to provide a substantial intake of dietary fiber through a variety of plant-based foods, including whole grains, legumes, fruits, vegetables, nuts, and seeds. Meals will be delivered bi-weekly, and compliance will be monitored through regular check-ins with a study dietitian.

SUMMARY:
This study aims to investigate the impact of various healthy diets, specifically a modified plant-based Mediterranean diet, on the gut microbiome and overall well-being post-colonoscopy. The investigators hypothesize that certain diets can positively influence gut bacteria, reducing inflammation and enhancing metabolic signals.

To explore this, they will utilize metagenomic testing on stool samples to analyze the DNA of gut microorganisms. Additionally, they will conduct immune profiling on serum samples and perform metabolomic analysis to comprehensively evaluate the diet-induced changes in immune response and metabolic pathways. This multi-faceted approach will help them understand how dietary changes affect the composition and function of the gut microbiome, immune function, and overall metabolism.

DETAILED DESCRIPTION:
An altered intestinal gut microbiota, i.e. dysbiosis, has been associated with the development of intestinal diseases including inflammatory bowel disease, colorectal cancer (CRC), and metabolic diseases such as obesity, type 2 diabetes mellitus (T2DM), and cardiovascular disease. Metagenomic analyses have revealed microbial biomarkers and ecological signatures in the fecal microbiome of CRC patients, correlating with chronic inflammation and gut dysbiosis. These factors have demonstrated prognostic relevance for CRC akin to other precursors, including conventional adenoma and serrated polyps.

Bowel lavage, a standard practice for facilitating colonoscopies, may affect the interaction between gut microbes and intestinal phenotypes. Standard bowel preparations have immediate impacts on gut microbiota composition, with alterations typically lasting around 14 days before a partial return to baseline. These changes in gut microbial diversity likely contribute to minor colonoscopy complications such as abdominal discomfort, bloating, diarrhea, and constipation during the recovery period.

Post-bowel lavage dietary intervention could potentially minimize lavage-associated side effects by promoting microbial diversity restoration and systemic inflammation reduction. In a previous mouse study, the investigators discovered that the Standard American Diet (SAD) led to the proliferation of opportunistic pathogens following surgical lavage. This change in microbial composition was linked to increased systemic inflammation and a higher incidence of surgical complications. Additionally, they observed that a high-fiber, low-saturated-fat diet-like a whole food, plant-based (WFPB), Med/DASH diet, and modified Mediterranean diet-can reverse this inflammatory phenotype.

However, there is a lack of interventional trials investigating the health benefits of specific dietary interventions following bowel lavage. Therefore, the investigators propose a human intervention study to assess if daily consumption of a high-fiber diet after colonoscopy will alter the intestinal microbiota, decrease inflammation, and improve digestive health.

This will be a controlled intervention study involving 30 subjects who will be enrolled on a rolling basis as they are identified during the recruitment period. The study begins with an initial visit at Week 1, where blood is collected for immune profiling and metabolomics, and participants start weekly stool collection using the S-Wipe method. At Week 2, a GutLab device is installed in participants' homes for daily stool collection. The colonoscopy occurs at Week 4, followed by a 2-week high-fiber diet provided by Thistle. Throughout the study, blood draws (6 mL) are performed at Weeks 1, 4, 6, and 8, while stool samples are collected weekly via S-Wipe and daily via GutLab. Participants log their food intake with a dietitian three times per week during Weeks 3, 5, and 7, and body composition measurements are taken before the colonoscopy and at the final visit. The study aims to quantify how dietary intervention affects post-lavage microbiome, metabolome, and immune response through analysis of blood and stool samples. Optional follow-ups at 1, 3, and 5 years will assess polyp recurrence. This design enables a comprehensive assessment of a high-fiber diet's impact on intestinal microbiota, inflammation, and digestive health in individuals with a history of polyps undergoing colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Due for 2nd or 3rd colonoscopy with prior diagnosis of tubular, villous, or serrated polyps but no current diagnosis of CRC.

Exclusion Criteria:

1. Inability to provide informed consent and engage in informed consent procedures.
2. Participants who suffer from allergic reactions to, or are unwilling to consume, any components of the dietary intervention.
3. Pregnant
4. Serious illness and in hospice or palliative care for terminal disease
5. Swallowing issues, including self-reported difficulty tolerating solids or liquids.
6. Active antibiotics use for an ongoing acute infection.
7. Any disorder, unwillingness, or inability not covered by any other exclusion criteria which, in the investigator's and/or team's opinion jeopardizes the safety of the participant or others or would interfere with adherence to the protocol.
8. Participants who plan to relocate to an area not served by UCSD or travel plans that do not permit completion of the study.
9. Possible ethanol (alcohol) use disorder defined by Alcohol Use Disorders Identification Test (AUDIT) score of >15

   Uncontrolled disease states:
10. Hyper-tension >160/100mmHg
11. Exacerbation of underlying gastrointestinal disease, including chronic inflammatory bowel disease or other malabsorptive disorders
12. Decompensated cirrhosis
13. Previously diagnosed Diabetes Mellitus with HbA1c >9% at screening
14. Newly diagnosed diabetes within the past three months, or HbA1c >6.5% at screening in a person not previously diagnosed with diabetes.
15. Participants with a history of end-stage renal disease (ESRD) on hemodialysis
16. Active infectious diseases (e.g., active tuberculosis < 3 months from symptom onset or positive test, COVID < 1 month from symptom onset or positive test)
17. Participants who require dietary restrictions due to a medical condition or are on a prescribed diet for underlying chronic diseases.
18. Participants with Type 1 or Type 2 diabetes on insulin
19. Participants aged 2: 75 years with Type 2 diabetes taking prescribed medications that can cause hypoglycemia (e.g., sulfonylureas, glinides), or on a prescribed diet
20. Hospitalization for a chronic disease (e.g., congestive heart failure, stroke) within the past three months
21. Requiring transfusions/apheresis during study period
22. Participants with a current diagnosis of, or who have received treatment for, bulimia or anorexia nervosa within the past 3 years
23. Participants with major psychiatric disorders, including major depression, schizophrenia, or psychosis, who have been hospitalized in the past six (6) months or are currently enrolled in treatment programs.
24. Hemoglobin <9.5 g/dL at screening
25. Myocardial infarction, invasive cardiac procedure, participation in a cardiac or acute rehabilitation programs, transient ischemic attacks, or unstable arrhythmias within the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Inflammatory Markers and Microbial Metabolites | 4 time-points throughout the study: Weeks 1, 4, 6, and 8
  Measure changes in circulating inflammatory markers (e.g., CRP, IL-6, IL-8, IL-10) and microbial metabolites (e.g., short-chain fatty acids such as butyrate, propionate, and acetate) at four time-points (Weeks 1, 4, 6, and 8) following bowel lavage and adherence to a modified plant-based Mediterranean diet. Gastrointestinal discomfort will be tracked using patient-reported outcome tools, with comparisons to baseline and across all time points.

SECONDARY OUTCOMES:
Changes in Gut Microbiome Composition and Opportunistic Pathogen Abundance | 7 Weeks of fecal sampling: Weeks 2-8
  Measure changes in the gut microbiome composition, including alpha diversity (e.g., Shannon index, Simpson index) and beta diversity (e.g., Bray-Curtis dissimilarity, UniFrac distances), along with the abundance of opportunistic pathogens (e.g., Enterococcus faecalis). Associations will be drawn between microbial diversity and composition, colonoscopy outcomes, circulating immune/metabolite markers, and reported gastrointestinal discomfort. Daily fecal samples will undergo metagenomic sequencing and bioinformatic analysis to quantify these metrics over 7 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego Altman Clinical and Translational Research Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code